CLINICAL TRIAL: NCT04686227
Title: Prevalence of Uterine Malformations in Newly Married Unselected Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sezcan Mumusoglu, Associate Professor, Hacettepe University
Other Study IDs: HU3643
Record Dates: First submitted 2020-12-18; First posted 2020-12-28 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Infertility
Keywords: Uterine Malformations; Fertility; Infertility; Pregnancy; Miscarriage
MeSH Terms: conditions — Infertility; Uterine Anomalies; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group-1, women with normal uterus
  Interventions: Diagnostic Test: 3D Ultrasound
- Group-2, women with any uterine malformations: Group-2 is going to be sub-grouped according to ASRM and ESHRE classifications
  Interventions: Diagnostic Test: 3D Ultrasound

INTERVENTIONS:
Diagnostic Test: 3D Ultrasound — Newly married women between the ages of 18-40 will be evaluated by 3D ultrasonography about the uterine morphology

SUMMARY:
Uterine malformation is occur due to the abnormal development of Mullerian canal during embryogenesis and it is known that it reduces the fertility and live birth rate and also increases the abortion and preterm birth rate. There are different classification methods have been used for defining the uterine malformations. The most common used classification method in the World is American Society of Reproductive Medicine (ASRM)'s system. In addition European Society of Human Reproduction and Embryology (ESHRE) and European Society for Gynaecological Endoscopy (ESGE) developed a new classification system. ASRM Uterine malformation Classification which is used for diagnosis and treatment of uterine malformations in our clinic is subdivided into 7 titles:

1. Agenesis or Hypoplasia -(a. Vaginal b. Cervical c. Fundal d. Tubal e. Combine)
2. Unicornuate -(a. Communicating Horn b. Non-Communicating Horn c. No Cavity d. No Horn)
3. Uterus Didelphus
4. Bicornuate Uterus-(a. Complete b. Partial)
5. Uterine Septum- (a. Complete b. Partial)
6. Arcuate Uterus
7. Diethylstilboestrol (DES) Related

The diagnosis of some of the uterine malformations have been done by using two dimensional (2D) ultrasonography, hysterosalphingography or surgically (laparoscopy or laparotomy) traditionally. A non-invasive procedure is required for the diagnosis of the uterine malformation, which is evaluating both the uterine contour and endometrial cavity.

In recent years frequently used three dimensional (3D) ultrasound is a non-invasive and quick diagnostic technique, and also it is sensitive as MRI. In hospital based case control studies, the frequency of uterine malformation was generally around 6%, while it was 8% in infertile patients and 12% in patients with abortion. However, there is a lack of prospective studies investigating the prevalence of uterine anomalies, fertility potential and effects on pregnancy outcomes in unselected patient groups in the literature. Therefore, at the high level evidence, there is no evidence that these anomalies affect fertility and pregnancy outcomes and should be corrected. In this study it was aimed to investigate the effects of uterine malformations on fecundability and pregnancy outcomes by evaluating the uterine morphology with 3D ultrasonography and calling for control purposes at the 1st and 2nd years of newly married women between the ages of 18-40.

DETAILED DESCRIPTION:
This study is designed as a prospective observational study. As it was mentioned above, it was aimed to investigate the effects of uterine malformations on fecundability and pregnancy outcomes by evaluating the uterine morphology with 3D ultrasonography and calling for control purposes at the 1st and 2nd years of newly married women between the ages of 18-40. Firstly a template flyer's designed to call the newly married women to our study. To be able to explain the study and call the participants officially, official permission's got from the municipal leading the wedding hall nearby the hospital (In Turkey, wedding halls are managed by the municipality covering their locations. As it's needed, the document can be added.). A scholarship student will explain the study and invite the couples. First and second year After the ultrasound, the participants will be called by phone to ask unprotected sex period; if conceived, outcomes of pregnancy (miscarriage, preterm birth, term birth, malpresentation etc.). Then the data will be worked on SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Husband is under 45 years old

Exclusion Criteria:

* Azospermia
* Women with Premature Ovarian Failure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Newly married women between the ages of 18-40
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of uterine malformations | 1 year after inclusion of last participant
  prevalence of uterine malformations in study population according to ASRM/ESHRE classifications
spontaneous fecundability | 1 year after inclusion of last participant
  1 year fecundability rate in subgroup of malformations and normal uterus
Pregnancy outcomes | During the pregnancy
  Rate of miscarriage, preterm birth, and malpresentation
Live birth rate | 1 year
  Having a live birth in all subgroups of uterine malformations and normal uterus
comparing of infertility rates | 1 year
  comparing of infertility rates between normal uterus population and every subgroup of uterine malformations

CONTACTS AND LOCATIONS:
Overall Officials: Sezcan Mumusoglu, Assoc. Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe UniversityHacettepe University School of Medicine, Department of Ob/Gyn, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Chan YY, Jayaprakasan K, Tan A, Thornton JG, Coomarasamy A, Raine-Fenning NJ. Reproductive outcomes in women with congenital uterine anomalies: a systematic review. Ultrasound Obstet Gynecol. 2011 Oct;38(4):371-82. doi: 10.1002/uog.10056. PMID 21830244
- [Background] Raga F, Bauset C, Remohi J, Bonilla-Musoles F, Simon C, Pellicer A. Reproductive impact of congenital Mullerian anomalies. Hum Reprod. 1997 Oct;12(10):2277-81. doi: 10.1093/humrep/12.10.2277. PMID 9402295
- [Background] Rackow BW, Arici A. Reproductive performance of women with mullerian anomalies. Curr Opin Obstet Gynecol. 2007 Jun;19(3):229-37. doi: 10.1097/GCO.0b013e32814b0649. PMID 17495638
- [Background] Tomazevic T, Ban-Frangez H, Ribic-Pucelj M, Premru-Srsen T, Verdenik I. Small uterine septum is an important risk variable for preterm birth. Eur J Obstet Gynecol Reprod Biol. 2007 Dec;135(2):154-7. doi: 10.1016/j.ejogrb.2006.12.001. Epub 2006 Dec 19. PMID 17182166
- [Background] Graupera B, Pascual MA, Hereter L, Browne JL, Ubeda B, Rodriguez I, Pedrero C. Accuracy of three-dimensional ultrasound compared with magnetic resonance imaging in diagnosis of Mullerian duct anomalies using ESHRE-ESGE consensus on the classification of congenital anomalies of the female genital tract. Ultrasound Obstet Gynecol. 2015 Nov;46(5):616-22. doi: 10.1002/uog.14825. Epub 2015 Oct 5. PMID 25690307
- [Background] Practice Committee of the American Society for Reproductive Medicine. Electronic address: ASRM@asrm.org; Practice Committee of the American Society for Reproductive Medicine. Uterine septum: a guideline. Fertil Steril. 2016 Sep 1;106(3):530-40. doi: 10.1016/j.fertnstert.2016.05.014. Epub 2016 May 25. PMID 27235766